CLINICAL TRIAL: NCT00622778
Title: Diagnostic Algorithm in Minor Head Injury
Brief Title: Immunemodulation in Patients With Minor Head Injury
Acronym: MHI
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Harald Wolf, Department for Trauma Surgery
Other Study IDs: 3-Wolf
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2011-07

CONDITIONS: Head Trauma
Keywords: intracranial bleeding; computed tomography scan
MeSH Terms: conditions — Craniocerebral Trauma; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum from peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients from daily practice

SUMMARY:
The purpose of this study is to try to prove the worth of the two (2) Serum Proteins S-100 Beta and NSE in combination with a diagnostic algorithm to help to establish diagnosis in patients with minor head injury.

ELIGIBILITY:
Inclusion Criteria:

* minor head injury

Exclusion Criteria:

* severe head injury

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from daily practice
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Intracranial Haematoma | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vilmos Vecsei, M.D. Professor, Study Chair — Head of Department
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Pelinka LE, Toegel E, Mauritz W, Redl H. Serum S 100 B: a marker of brain damage in traumatic brain injury with and without multiple trauma. Shock. 2003 Mar;19(3):195-200. doi: 10.1097/00024382-200303000-00001. PMID 12630517
- [Background] Pelinka LE, Bahrami S, Szalay L, Umar F, Redl H. Hemorrhagic shock induces an S 100 B increase associated with shock severity. Shock. 2003 May;19(5):422-6. doi: 10.1097/01.shk.0000055345.58165.52. PMID 12744484
- [Background] Pelinka LE, Kroepfl A, Leixnering M, Buchinger W, Raabe A, Redl H. GFAP versus S100B in serum after traumatic brain injury: relationship to brain damage and outcome. J Neurotrauma. 2004 Nov;21(11):1553-61. doi: 10.1089/neu.2004.21.1553. PMID 15684648
- [Derived] Wolf H, Frantal S, Pajenda GS, Salameh O, Widhalm H, Hajdu S, Sarahrudi K. Predictive value of neuromarkers supported by a set of clinical criteria in patients with mild traumatic brain injury: S100B protein and neuron-specific enolase on trial: clinical article. J Neurosurg. 2013 Jun;118(6):1298-303. doi: 10.3171/2013.1.JNS121181. Epub 2013 Mar 1. PMID 23451906